CLINICAL TRIAL: NCT05084547
Title: A Comparison of Upper Extremity Exercise Capacity and Activities of Daily Living Between Subjects With Bronchiectasis and Healthy Controls
Brief Title: Comparison of Upper Extremity Exercise Capacity and ADL Between Subjects With Bronchiectasis and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Research Assistant, Hacettepe University
Other Study IDs: GO 20/55
Record Dates: First submitted 2021-09-29; First posted 2021-10-20 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Subjects with Bronchiectasis
  Interventions: Other: No intervention
- Control: Healthy Controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Bronchiectasis is a chronic lung disease characterized by permanent dilatation and destruction, resulting from the destruction of elastic tissue and muscular components in the bronchial walls, due to infection or inflammation. The exercise tolerance, physical activity level, respiratory and peripheral muscle strength of patients with bronchiectasis are lower than those of healthy individuals. The decrease in exercise tolerance occurs while performing upper extremity activities as well as lower extremity tasks. Many studies have reported that upper extremity exercise capacity is reduced in chronic obstructive pulmonary disease (COPD), a disease similar to bronchiectasis, and that patients often experience significant dyspnea and fatigue during upper extremity tasks that are important for daily life. The mechanisms causing this situation may be neuromechanical dysfunction of the respiratory muscles (diaphragm and accessory respiratory muscles) (thoracoabdominal asynchrony) and changes in lung volume in activities involving the upper extremities. The disturbances in ventilatory mechanics in patients with COPD cause upper extremity exercise to be terminated at low workloads compared to healthy individuals. Upper extremity exercise has been defined as part of pulmonary rehabilitation. The determination of upper extremity exercise capacity may play a predictive role in maintaining and improving upper extremity and daily life activity level in patients with chronic lung disease.

Six-minute Pegboard and Ring test (6PBRT) is used to evaluate extremity exercise capacity and upper extremity function and endurance. The 6PBRT score and upper extremity daily living activities show a clear relationship in patients with COPD, and it can be used to determine and improve the performance of daily living activities in pulmonary rehabilitation programs. Glittre Activities of Daily Living (Glittre ADL test) covers activities that are necessary for daily living and commonly used activities. The Glittre ADL test produces similar cardiorespiratory responses when compared with the six-minute walk test. In this study, unsupported upper extremity exercise capacity and upper extremity function/endurance and the performance of daily living activities will be compared in participants with bronchiectasis and compared with healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bronchiectasis and being clinically stable,
* Being 18 years old or older,
* Being able and willing to complete the informed consent process.

Exclusion criteria:

* Individuals with bronchiectasis whose clinical condition is unstable,
* Individuals with bronchiectasis who have severe neuromuscular, musculoskeletal, and rheumatological problems,
* Being unable to cooperate,
* Not being willing to participate in the study

The healthy controls will be composed of individuals who volunteered for the study without any known disease. Healthy individuals who did not volunteer to participate in the study will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with bronchiectasis and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test - Forced vital capacity | 1st day
  Pulmonary function test using a spirometer will be performed. Forced vital capacity will be recorded.
Pulmonary function test - Forced expiratory volume in one second | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second will be recorded.
Pulmonary function test - Forced expiratory volume in one second/Forced vital capacity | 1st day
  Pulmonary function test using a spirometer will be performed. Forced expiratory volume in one second/Forced vital capacity in one second will be recorded.
Pulmonary function test - Peak expiratory flow | 1st day
  Pulmonary function test using a spirometer will be performed. Peak expiratory flow will be recorded.
Pulmonary function test - Forced mid-expiratory flow (FEF25-75) | 1st day
  Pulmonary function test using a spirometer will be performed. Forced mid-expiratory flow (FEF25-75) will be recorded.
Glittre Activities of Daily Living Test | 1st day
  The test covers activities that are necessary for daily living and commonly used activities that are known to be difficult for patients with COPD.
Unsupported upper extremity exercise capacity | 1st day
  Upper extremity exercise capacity will be evaluated using 6PBRT. During the test, the patient is asked to sit in front of a pegboard and move as many rings as possible from the two lower holes to the two upper holes, using both hands simultaneously, for six minutes. The number of rings carried during the six minutes constitutes the final score. Heart rate and oxygen saturation with pulse oximetry before and after the test, dyspnea, arm and general fatigue will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Aslihan Cakmak, MSc, Study Director — Hacettepe University; Deniz Inal-Ince, PhD, Study Chair — Hacettepe University; Lutfi Coplu, MD, Principal Investigator — Hacettepe University; Hazal Sonbahar-Ulu, PhD, Principal Investigator — Akdeniz University; Ebru Calik-Kutukcu, PhD, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, PhD, Principal Investigator — Hacettepe University; Melda Saglam, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cakmak A, Kocaaga E, Sonbahar-Ulu H, Inal-Ince D, Vardar-Yagli N, Calik-Kutukcu E, Saglam M, Coplu L. Upper Extremity Exercise Capacity and Activities of Daily Living in Individuals With Bronchiectasis Versus Healthy Controls. Phys Ther. 2023 Apr 4;103(4):pzad012. doi: 10.1093/ptj/pzad012. PMID 37086209